CLINICAL TRIAL: NCT05305690
Title: Natural History and Nonoperative Management of Penetrating Cerebrovascular Injury
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Poudre Valley Health System (Other)
Collaborators: Denver Health Medical Center (Other)
Responsible Party: Principal Investigator, Cordelie Witt, Investigator, Poudre Valley Health System
Other Study IDs: 19-0647
Record Dates: First submitted 2022-02-25; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Cerebrovascular Trauma
Keywords: penetrating cerebrovascular injury; nonoperative management; penetrating neck trauma; natural history; antithrombotic therapy; case series
MeSH Terms: conditions — Cerebrovascular Trauma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Penetrating cerebrovascular injury, managed nonoperatively: PCVI from penetrating trauma without upfront operation
  Interventions: Other: No intervention
- Penetrating cerebrovascular injury, managed operatively
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This study did is a retrospective case series and does not involve an intervention. Investigators will compare patients managed operatively vs nonoperatively, focused on nonoperative therapy.

SUMMARY:
The goal of this study is to evaluate a series of cases of penetrating cerebrovascular injury managed without upfront operation. Investigators focus on patient characteristics, injury details, treatment modalities, serial imaging studies, patient outcomes, and complications. Investigators will compare this patient population to patients managed with upfront operation for context.

DETAILED DESCRIPTION:
Penetrating cerebrovascular injuries (PCVIs) are uncommon, with little data to guide management when emergent operative repair is not performed. Investigators hypothesized that PCVIs may be managed with antithrombotic therapy and directed use of endovascular interventions, but that PCVIs may require enhanced surveillance due to a risk of delayed complications. To perform this study, investigators will review patients with penetrating carotid and vertebral artery injuries managed at an urban Level I trauma center from 2016 to 2022. Patients will be included if they underwent initial nonoperative management (NOM). Patient characteristics, injury details, treatments, serial imaging, outcomes, and complications will be assessed in a retrospective manner using chart abstraction. Investigators will briefly compare these patients to those managed with upfront operations for context.

ELIGIBILITY:
Inclusion Criteria:

* Penetrating neck trauma
* Carotid or vertebral artery injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators are including all adult patients with penetrating cerebrovascular injury since 5/1/2016 to present. Investigators will focus on those managed without operative intervention, but will include cases managed operatively for comparison.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2023-01-03 (Estimated); Study Completion 2023-01-03 (Estimated)

PRIMARY OUTCOMES:
number of patients with stroke | up to one year post-injury
  ischemic stroke

SECONDARY OUTCOMES:
number of patients with injury progression | up to one year post-injury
  CTA progression of PCVI severity (Grade)
number of patients with death | up to one year post-injury
  death
number of patients with bleeding complications | up to one year post-injury
  intracranial hemorrhage, GI bleed, etc requiring change in treatment
number of patients treated with operative exploration | up to one year post-injury
  All patients in cohort are treated with initial trial of nonoperative management. This outcome assesses the number of patients who subsequently required operative neck exploration. This is readily attainable from operative reports.
number of patients treated with arterial embolization or arterial stent placement | up to one year post-injury
  IR procedures are adjuncts to nonoperative management. Performance of these procedures is readily attainable from IR procedure reports.

IPD SHARING:
Plan to Share IPD: No
Data is not readily sharable due to HIPAA restrictions